CLINICAL TRIAL: NCT00733018
Title: Health Risk Assessment of Dietary Carbohydrates in Chronic Disease Development
Brief Title: Nutrigenomics Diet Intervention Study Comparing Effects of Western and Balanced Diet in Healthy Subjects
Acronym: Foodgene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); FUGE Mid-Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: REK 4.2007.515; 16649 (Other: NSD)
Record Dates: First submitted 2008-08-11; First posted 2008-08-12 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Cardiovascular Diseases; Chronic Disease
Keywords: Nutrigenomics; Gene Expression; Diet, Carbohydrate-Restricted; Life Style; Health Behavior
MeSH Terms: conditions — Cardiovascular Diseases; Chronic Disease; Health Behavior | interventions — Diet, Western; Diet, Fat-Restricted; Diet, Protein-Restricted; Diet, High-Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Diet A - Western diet
  Interventions: Behavioral: "Western" versus "balanced" macro nutrient diet composition
- B (Active Comparator): Diet B - Balanced diet
  Interventions: Behavioral: "Western" versus "balanced" macro nutrient diet composition

INTERVENTIONS:
Behavioral: "Western" versus "balanced" macro nutrient diet composition — Randomized crossover diet intervention. 6 days on solely one of two isocaloric diets, 8 days washout, and then the other diet for 6 days. Fasting blood sampling before and after each diet intervention period.
  Other Names: western diet; high-carbohydrate, low fat, low protein diet; balanced diet; low-carbohydrate, high fat, high protein diet

SUMMARY:
Diet macronutrient relative composition, quality and quantity determines lifestyle disease, including cardiovascular disease, development. Our hypothesis is that a high content of carbohydrates in the diet contributes to increased insulin level. Moreover, activating enzymes promoting inflammatory processes and possibly chronic disease development in the body.

DETAILED DESCRIPTION:
The most frequent cause of death in both women and men in the western world is cardiovascular artery disease (CAD). Well accepted as a lifestyle disease, known risk factors for CAD development include changes in blood lipid content and type as well as micro inflammation in the arterial wall. Low density lipoprotein (LDL) and triglycerides are increased, high density lipoprotein (HDL) is reduced. Furthermore, type II diabetes, metabolic syndrome, hypertension, overweight, reduced physical activity and smoking also precede CAD development. Common for many of the risk factors is that they are induced by improper diet. Recent research has shown that especially total amount, composition and quality of the macro nutrients, protein, carbohydrate and fats, is important. In this project we will explore changes in blood gene expression in response to a western and a balanced crossover diet intervention.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* BMI 24.5-27.5
* pass health check criteria

Exclusion Criteria:

* chronic diseases
* inflammation
* pregnancy and lactation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Changes in microarray gene expression profiles in blood from healthy young women and men, in response to western or balanced dietary macro nutrient composition. | Before and after each of two 6-days diet intervention periods

SECONDARY OUTCOMES:
Inflammatory markers, hormonal dietary responses and blood lipids | Before and after each of two 6-days diet intervention periods

CONTACTS AND LOCATIONS:
Overall Officials: Berit Johansen, PhD, Principal Investigator — Norwegian University of Sciense and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Background] Brattbakk HR, Arbo I, Aagaard S, Lindseth I, de Soysa AK, Langaas M, Kulseng B, Lindberg F, Johansen B. Balanced caloric macronutrient composition downregulates immunological gene expression in human blood cells-adipose tissue diverges. OMICS. 2013 Jan;17(1):41-52. doi: 10.1089/omi.2010.0124. Epub 2011 Jun 16. PMID 21679058